CLINICAL TRIAL: NCT01193049
Title: A Two-Part, Randomized Clinical Trial to Study the Effects of a Single Dose of Prednisone on Biomarkers of Allergen Responses in Asthmatics
Brief Title: A Study on the Effects of a Single Dose of Prednisone on Biomarkers of Allergen Responses in Asthmatics (MK-0000-175)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000-175; 2010-020518-27 (EudraCT Number: From the European Union Drug Regulatory Authorities Clinical Trial System)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2012-08-02 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Asthma
Keywords: Nasal Allergen Challenge, Inhaled Allergen Challenge, Asthma
MeSH Terms: conditions — Asthma | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone, then Placebo (Experimental): Prednisone in the first crossover treatment period and placebo in the second crossover treatment period
  Interventions: Drug: Prednisone; Drug: Placebo
- Placebo, then Prednisone (Experimental): Placebo in the first crossover treatment period and prednisone in the second crossover treatment period
  Interventions: Drug: Prednisone; Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Prednisone (25 mg) tablets as a single oral dose on Day 1 of each study period
Drug: Placebo — Matching placebo tablets as a single oral dose on Day 1 of each study period

SUMMARY:
The purpose of this study is to evaluate the relationship between upper and lower airway allergen-induced cytokine responses in mild asthmatics by attempting to demonstrate the following: 1) a positive correlation between allergen-induced Type 2 T-helper cell (Th2) cytokines (interleukins 5 and 13) in sputum and nasal exudates; and 2) a positive correlation between effects of prednisone versus placebo on Th2 cytokines in sputum and nasal exudates.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical history of mild to moderate asthma for at least 6 months, but otherwise is in good health
* Participant with allergic rhinitis and asthma has a history of nonseasonal airway symptoms in response to aeroallergens OR has seasonal symptoms but can be evaluated out-of-season
* Is clinically stable and free of respiratory infection or change in allergen exposure for at least 4 weeks prior to start of study

Exclusion Criteria:

* Has intolerance to the study drug, inhaled salbutamol, antihistamines, or any other potential asthma/anaphylaxis rescue medication
* Has intolerance to lidocaine/lignocaine, sedatives, atropine or glycopyrrolate, or any other medication associated with bronchoscopy
* Has taken oral parenteral corticosteroids within 8 weeks or inhaled corticosteroids/nasal corticosteroids within 5 weeks of screening and/or during the study
* Has recent (4 weeks) or ongoing upper or lower respiratory tract infection
* Has active allergic rhinitis at screening
* Has received a vaccination within 3 weeks of screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone, Then Placebo: Prednisone in the first double blind treatment period and placebo in the second double blind treatment period
- Placebo, Then Prednisone: Placebo in the first double blind treatment period and prednisone in the second double blind treatment period
Period: Period 1: Placebo Run-In
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Washout 1 : 21 Day Washout
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Period 2 : Double Blind Crossover
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Washout 2 : 21 Day Washout
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Period 3 : Double Blind Crossover
Arm/Group | Prednisone, Then Placebo | Placebo, Then Prednisone
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Change From Baseline in Interleukin-5 (IL-5) Concentration From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, nasal exudates (NE) and sputum (SP) were collected, then the concentrations of IL-5 were determined from NE and SP collected after 7 hours and previously at baseline (BL), to derive the fold change (FC) from BL for each participant. The geometric mean (GM) was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Groups:
- Prednisone: All participants who received at least one dose of prednisone
- Placebo: All participants who received at least one dose of placebo
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  Sputum | 2.16 [1.25 to 3.74] | 8.60 [3.82 to 19.34]
  Nasal Exudate | 1.69 [0.88 to 3.26] | 8.63 [4.45 to 16.77]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM Fold Reduction (FR) is the GM of individual FC(Prednisone)/FC (Placebo) from SP; Test type: Superiority or Other; p = 0.001, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: SP = 0.25, 90% CI 2-sided [0.14 to 0.46]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR is the GM of individual FC(Prednisone)/FC(Placebo) from NE; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided p value, α = 0.05; GM FR from Placebo : NE = 0.20, 90% CI 2-sided [0.13 to 0.30]
Statistical Analysis 3: Comparison: Placebo; Correlation between SP and NE of FC from BL in IL-5 after placebo treatment; Test type: Superiority or Other; p = 0.553, Pearson's correlation coefficient — Unadjusted for Baseline and Period Effects; Correlation FC from BL: SP vs NE = 0.20
Statistical Analysis 4: Comparison: Prednisone; Correlation between SP and NE of FR from placebo in IL-5 after prednisone treatment; Test type: Superiority or Other; p = 0.964, Pearson's correlation coefficient — Unadjusted for Baseline and Period Effects; Correlation FR from Placebo :SP vs NE = -0.02

2. Primary Outcome: Geometric Mean Fold Change From Baseline in Interleukin-13 (IL-13) From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of IL-13 were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  Sputum | 1.57 [1.21 to 2.04] | 5.86 [2.57 to 13.36]
  Nasal Exudate | 1.02 [0.65 to 1.58] | 3.29 [1.82 to 5.95]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM FR is the GM of individual FC(Prednisone)/FC (Placebo) from SP; Test type: Superiority or Other; p = 0.009, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: SP = 0.27, 90% CI 2-sided [0.12 to 0.62]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR is the GM of individual FC Prednisone)/FC(Placebo) from NE; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo : NE = 0.31, 90% CI 2-sided [0.22 to 0.43]
Statistical Analysis 3: Comparison: Placebo; Correlation between SP and NE of FC from BL in IL-13 after placebo treatment; Test type: Superiority or Other; p = 0.962, Pearson's correlation coefficient — Unadjusted for Baseline and Period Effects; Correlation FC from BL: SP vs NE = -0.02
Statistical Analysis 4: Comparison: Prednisone; Correlation between SP and NE of FR from placebo in IL-13 after prednisone treatment; Test type: Superiority or Other; p = 0.83, Pearson's correlation coefficient — Unadjusted for Baseline and Period Effects; Correlation FR from Placebo: SP vs NE = 0.07

3. Secondary Outcome: Geometric Mean Fold Change From Baseline in Thymus and Activation Regulated Chemokine (TARC) From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of TARC were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  Sputum | 1.63 [1.22 to 2.17] | 2.04 [1.21 to 3.46]
  Nasal Exudates | 1.33 [0.88 to 2.01] | 1.22 [0.96 to 1.57]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) from SP; Test type: Superiority or Other; p = 0.258, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: SP = 0.80, 90% CI 2-sided [0.43 to 1.47]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) from NE; Test type: Superiority or Other; p = 0.681, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: NE = 1.08, 90% CI 2-sided [0.80 to 1.46]

4. Secondary Outcome: Geometric Mean Fold Change From Baseline in Eotaxin-3 From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of Eotaxin-3 were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  Sputum | 1.30 [0.67 to 2.51] | 2.14 [1.41 to 3.24]
  Nasal Exudates | 0.86 [0.56 to 1.31] | 1.35 [0.66 to 2.74]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) from SP; Test type: Superiority or Other; p = 0.117, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo:SP = 0.61, 90% CI 2-sided [0.30 to 1.24]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) from NE; Test type: Superiority or Other; p = 0.011, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: NE = 0.64, 90% CI 2-sided [0.47 to 0.86]

5. Secondary Outcome: Change in Vibration Response Imaging (VRI) After Metacholine Exposure
Description: One hour before treatment with prednisone/placebo, participants inhaled for 2 minutes a nebulised solution of metacholine (0.13 ml/min); then one hour after prednisone/placebo treatment were challenged with allergens. From 1 to 7 hours after allergen challenge, ventilatory heterogeneity was assessed by Vibration Response Imaging (VRI) by monitoring the following: inspiration/expiration (I/E) amplitude ratio, I/E duration ratio, synchrony duration, and quantitative lung data.
Time Frame: From 1 to 7 hours post-allergen challenge
Population: As all VRI results showed no allergen or treatment-related signals these results are not presented.
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Geometric Mean Fold Change From Baseline in RNA Expression for Genes Encoding IL-5 and IL-13 From Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, SP were collected, then the RNA expression profiles of IL-5 and IL-13 genes were determined from SP collected after 7 hours and previously at baseline, to derive the FC from BL for each participant. The GM was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  IL-5 | 4.87 [3.20 to 7.39] | 7.37 [5.96 to 9.11]
  IL-13 | 2.90 [2.42 to 3.48] | 3.93 [3.02 to 5.13]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) for IL-5; Test type: Superiority or Other; p = 0.010, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: IL-5 = 1.51, 90% CI 2-sided [1.15 to 1.99]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC(Prednisone)/FC (Placebo) for IL-13; Test type: Superiority or Other; p = 0.020, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: IL-13 = 1.35, 90% CI 2-sided [1.07 to 1.71]

7. Secondary Outcome: Geometric Mean Fold Change From Baseline in Interleukin-17 (IL-17) From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of IL-17 were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  Sputum | 0.68 [0.58 to 0.80] | 0.83 [0.71 to 0.98]
  Nasal Exudates | 0.84 [0.48 to 1.46] | 1.23 [1.14 to 1.33]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) in IL-17 from SP; Test type: Superiority or Other; p = 0.119, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: SP = 0.82, 90% CI 2-sided [0.62 to 1.09]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) in IL-17 from NE; Test type: Superiority or Other; p = 0.103, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: NE = 0.68, 90% CI 2-sided [0.41 to 1.14]

8. Secondary Outcome: Geometric Mean Fold Change From Baseline in Interleukin-1β (IL-1β) From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of IL-1β were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  Sputum | 0.80 [0.55 to 1.17] | 1.34 [0.86 to 2.09]
  Nasal Exudates | 0.19 [0.14 to 0.27] | 0.39 [0.24 to 0.63]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) in IL-1β from SP; Test type: Superiority or Other; p = 0.003, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: SP = 0.60, 90% CI 2-sided [0.46 to 0.77]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC(Prednisone)/FC (Placebo) in IL-1β from NE; Test type: Superiority or Other; p = 0.036, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: NE = 0.49, 90% CI 2-sided [0.26 to 0.93]

9. Secondary Outcome: Geometric Mean Fold Change From Baseline in Macrophage Inflammatory Protein-1β (MIP-1β) From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of MIP-1β were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: All randomized participants
Measure: Geometric Mean (90% Confidence Interval); unit: Fold Change
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 11 | 11
Fold Change
  Sputum | 1.35 [0.75 to 2.43] | 1.92 [0.94 to 3.93]
  Nasal Exudates | 0.73 [0.47 to 1.13] | 1.19 [0.70 to 2.01]
Statistical Analysis 1: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC(Prednisone)/FC (Placebo) in MIP-1β from SP; Test type: Superiority or Other; p = 0.143, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: SP = 0.70, 90% CI 2-sided [0.40 to 1.24]
Statistical Analysis 2: Comparison: Prednisone vs Placebo; GM FR from Placebo is the GM of individual FC (Prednisone)/FC (Placebo) in MIP-1β from NE; Test type: Superiority or Other; p = 0.056, ANOVA — 1-sided p-value, α = 0.05; GM FR from Placebo: NE = 0.61, 90% CI 2-sided [0.37 to 1.02]

10. Secondary Outcome: Geometric Mean Fold Change From Baseline in Thymic Stromal Lymphopoietin (TSLP) From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of TSLP were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was planned to be determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: As TSLP levels were too low to detect, this analysis was not performed and results are not presented.
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Geometric Mean Fold Change From Baseline in Interleukin-23 (IL-23) From Nasal Exudates and Sputum at 7 Hours Post-allergen Challenge
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then the concentrations of IL-23 were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was plan to be determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: As IL-23 levels were too low to detect, this analysis was not performed and results are not presented.
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Geometric Mean Fold Change From Baseline in Cytokines From Bronchoalveolar Lavage Fluid (BALf)
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 23 hours had elapsed, BALf were collected, then the concentrations of IL-5, IL-13, and TARC were determined from BALf collected after 23 hours and previously at BL, to derive the FC from BL for each participant. The GM was planned to be determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 23 hours post-allergen challenge
Population: As concentrations of cytokines were below the lower limit of quantitation this analysis was not performed, and results are not presented.
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Geometric Mean Fold Change From Baseline in Nasal and Bronchial Eicosanoids and Leukotrienes at 7 Hours Post-allergen Challenge.
Description: Participants were treated with either prednisone or placebo, followed 1 hour later by nasal allergen challenge and then inhaled allergen challenge. After 7 hours had elapsed, NE and SP were collected, then prostaglandin and leukotriene concentrations were determined from NE and SP collected after 7 hours and previously at BL, to derive the FC from BL for each participant. The GM was planned to be determined by averaging FC from BL for all analyzed participants.
Time Frame: Baseline and 7 hours post-allergen challenge
Population: As this same approach in a parallel study was unfruitful, these data were not pursued, and results are not presented.
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All participants in this crossover study received both prednisone and placebo.
Arm/Group | Prednisone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone (N=11) | Placebo (N=11)
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.